CLINICAL TRIAL: NCT03270787
Title: A Randomized, Double Blind, Placebo-controlled Study of Compound Danshen Dripping Pills in Preventing and Treating Acute Mountain Sickness
Brief Title: Study of Compound Danshen Dripping Pills to Treat Acute Mountain Sickness
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tasly Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCM1421
Record Dates: First submitted 2016-06-23; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Acute Mountain Sickness
Keywords: Acute Mountain sickness; Compound Danshen Dripping Pills
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Comparator (Placebo Comparator): Placebo Comparator: controlled group Placebo,10pills,tid,po
  Interventions: Drug: Placebo
- Compound danshen dripping pills (Experimental): Compound danshen dripping pills Compound danshen dripping pills ,10pills,tid,po
  Interventions: Drug: Compound danshen dripping pills

INTERVENTIONS:
Drug: Placebo — Drug: Placebo Placebo,10pills,tid,treat 1 weeks.
  Arms: Placebo Comparator
Drug: Compound danshen dripping pills — Drug: Compound danshen dripping pills Compound danshen dripping pills,10pills,tid,treat 1 weeks.
  Arms: Compound danshen dripping pills

SUMMARY:
This study is to evaluate the efficacy and safety of compound danshen dripping pills in preventing and treating acute mountain sickness.

DETAILED DESCRIPTION:
Compound danshen dripping pills is mainly used for the treatment and prevention of coronary heart disease and high-risk groups ,consists of Danshen (Radix Salviae Miltiorrhizae), Sanqi (Radix Notoginseng) and borneol.Danshen is the main drug efficacy of stasis, nourishing the nerves.Pharmacological studies have shown that Danshen can improve the oxygen carrying capacity of blood, increase oxygen supply to vital organs, effectively reduce hypoxia-induced heart and other vital organs, brain and kidney damage. Danshen can activate the fibrinolytic system, reduce blood viscosity, clear the microcirculation, promote blood circulation, increasing the amount of tissue oxygen by inhibiting platelet aggregation.This study is being conducted to evaluate the efficacy and safety of compound danshen dripping pills in preventing and treating acute mountain sickness, when compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-45 years，Male or female, plain natives
* first stationed at high altitude above 3,000 meters
* Upon physical examination before enrollment in good health
* BMI 19 to 24; (weight kg / height Sqm )
* voluntary signs the informed consent

Exclusion Criteria:

* menstruation, pregnancy and breast-feeding women
* smoking, alcohol and drug abusers
* Clear history of drug allergy or allergic persons
* application of various drugs (including traditional Chinese medicine) two weeks ago
* Combined with severe liver and kidney dysfunction (cardiac function Grade ≥3, liver function Grade > 2 times of the upper limit of normal, Cr> upper limit of normal);
* Subject with blood donation experiences or blood test experiences within three months before be selected.
* C- reactive protein test results exceed the upper limit of normal.
* clinically significant gastrointestinal disease, mental illness and diabetes, hyperthyroidism and other metabolic diseases;
* Past suffering from cardiovascular and cerebrovascular disease
* fatigue syndrome that is not by high altitude-induced
* primary headache
* Vomiting due to other causes, such as digestive disorders as a result of the vomiting reflex, vomiting vestibular disorders, neurotic vomiting;
* Allergies
* Who participated in clinical trials of other drugs within a month
* blood circulation, increase immunity and antioxidant drug users

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2016-06-24 (Actual); Primary Completion 2016-07-13 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
The incidence of acute mountain sickness rapid radical to an altitude of 3000m above the plateau region compared to placebo | 7days

CONTACTS AND LOCATIONS:
Overall Officials: Min Zhao, PhD, Study Director — Tasly Group, Co. Ltd.
Locations (1):
- People's Hospital of Tibet Autonomous Region, Damxung, Tibet, China

IPD SHARING:
Plan to Share IPD: No